CLINICAL TRIAL: NCT04557371
Title: A Clinical Study to Assess the Local Cutaneous and Ocular Tolerance of Three Developmental Cosmetic Facial Skin Care Formulations in Healthy Females With Clinically Assessed Sensitive Skin.
Brief Title: A Study to Assess the Local Cutaneous and Ocular Tolerance of Three Developmental Facial Skin-care Formulations.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 213059
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-02

CONDITIONS: Skin Care
Keywords: Glycerol; Niacinamide; Skin Care

STUDY DESIGN:
Intervention Model Description: The study is a randomized, 3-arm parallel group study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluator-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Developmental Serum (Experimental): The participants will apply a developmental serum topically to the face twice daily (morning and evening) to freshly cleansed with normal moisturizing routine for 21 days.
  Interventions: Other: Serum
- Developmental Lotion (Experimental): The participants will apply a developmental lotion topically to the face twice daily (morning and evening) to freshly cleansed skin for 21 days.
  Interventions: Other: Lotion
- Developmental Cream (Experimental): The participants will apply a developmental cream topically to the face twice daily (morning and evening) to freshly cleansed skin for 21 days.
  Interventions: Other: Cream

INTERVENTIONS:
Other: Serum — Participants will topically apply the serum to the face as per normal home use application in place of their current facial serum product.
  Arms: Developmental Serum
Other: Lotion — Participants will topically apply lotion to the face as per normal home use application in place of their current facial lotion product.
  Arms: Developmental Lotion
Other: Cream — Participants will topically apply cream to the face as per normal home use application in place of their current facial cream product.
  Arms: Developmental Cream

SUMMARY:
This study aims to determine the local cutaneous and ocular tolerance of 3 developmental skin-care products; a serum, a lotion, and a cream in healthy female subjects with clinically evaluated sensitive facial skin for 21 days.

DETAILED DESCRIPTION:
This will be a randomized, non-comparative, single-blind (evaluator), 3-arm, parallel-group, single-center, clinical 'in-use' study to determine the local cutaneous and ocular tolerance profiles of 3 developmental cosmetic facial skincare products; a serum, lotion, and cream in healthy females with clinically-evaluated sensitive skin as determined by a positive response to a Lactic Acid Stinging Test (LAST) with signs or symptoms of cutaneous irritation and no ophthalmological conditions. Assessments will be performed and recorded for 21 days.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, the application schedule, the lifestyle guidelines, and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee , no clinically significant/relevant abnormalities in medical history or upon dermatologist and ophthalmologist examination, or condition, that would impact the participant's safety, well-being or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participants with sensitive facial skin, defined as a positive response to a LAST in the nasolabial area.
* A participant with a dermatologist signs and symptoms of cutaneous irritation score of 0.5 (very slight) or greater for erythema per dermatological evaluation.
* A participant with a dermatologist signs and symptoms of cutaneous irritation score of 0.5 (very slight) or greater for dryness per dermatological evaluation.
* A participant with a dermatologist signs and symptoms of cutaneous irritation score of 0 (none) or 0.5 (very sight) for scaling per dermatological evaluation.
* A participant with a dermatologist signs and symptoms of cutaneous irritation score of 0 (none) or 0.5 (very sight) for edema per dermatological evaluation.
* A participant with an ophthalmologist total signs and symptoms of ocular irritation score of zero (0) per dermatological evaluation.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GSK CH employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant who is pregnant (self-reported) or intends to become pregnant during the study duration.
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the protocol lifestyle considerations required by this study, as described in this protocol.
* A participant with current or recent (within last 6 months before the start of the study) history of atopic lesions and/or eczema.
* A participant with a history of allergic reactions to topical-use products, cosmetics or medications or their ingredients.
* A participant with any history of significant diseases or medical conditions known to alter skin or eye appearance or physiologic response (e.g. diabetes) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction.
* A participant presenting open sores, pimples, or cysts at the application site (face).
* A participant considered immune-compromised.
* A participant who has used any of the following topical or systemic medications up to two weeks before the screening visit: immuno-suppressants, antihistamines, non-steroidal anti-inflammatory drugs (NSAIDS), and/or corticosteroids.
* A participant who has used oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit.
* A participant who has been vaccinated up to 1 month before the screening visit or who is intending to receive a vaccination during their participation in the study.
* A participant with a recent history (within the last 5 years) of alcohol or other substance abuse.
* A participant with any skin marks on the face that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles).
* A participant who has previously been enrolled in this study.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* Participants with corneal ulcers, keratoconus, blepharitis, meibomitis, pterygium, chemosis, moderately or severe hyperaemia or other active ocular diseases.
* A participant currently using any medication which in the opinion of the investigator (medically qualified designee) may affect the evaluation of the investigational product or place the participant at undue risk.
* A participant with an active dermatosis (local or disseminated) that might interfere with the results of the study.
* A participant with a dermatologist signs and symptoms of cutaneous irritation score of 3 (severe) for edema, scaling, erythema, or dryness per dermatological evaluation.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Schenefeld, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Germany.
Pre-assignment Details: A total of 286 participants were screened of which 150 participants were enrolled and allocated to a randomized treatment. A total of 147 participants completed the study.
Groups:
- Developmental Serum: The first topical application of the developmental serum was applied by the participants at the study site under the supervision of a trained technician. Participants were instructed to apply developmental serum at home again the same evening of their first supervised application and then twice daily for a total of 21 days, as part of their normal skin care routine. The final application of developmental serum was performed at home on the morning of the final visit.
- Developmental Lotion: The first topical application of the developmental lotion was applied by the participants at the study site under the supervision of a trained technician. Participants were instructed to apply developmental lotion at home again the same evening of their first supervised application and then twice daily for a total of 21 days, as part of their normal skin care routine. The final application of developmental lotion was performed at home on the morning of the final visit.
- Developmental Cream: The first topical application of the developmental cream was applied by the participants at the study site under the supervision of a trained technician. Participants were instructed to apply developmental cream at home again the same evening of their first supervised application and then twice daily for a total of 21 days, as part of their normal skin care routine. The final application of developmental cream was performed at home on the morning of the final visit.
Period: Overall Study
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Started | 50 | 49 | 51
Completed | 49 | 47 | 51
Not Completed | 1 | 2 | 0
Not completed — Covid-19-related | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population comprised of all randomized participants who had at least one application of the study product (serum, lotion, or cream)
Groups:
- Total: Total of all reporting groups
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream | Total
Number analyzed (Participants) | 50 | 49 | 51 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (11.06) | 47.8 (11.30) | 44.6 (13.72) | 47.0 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 51 | 150
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 3 | 0 | 0 | 3
  Asian - East Asian Heritage | 0 | 1 | 0 | 1
  Asian - South East Asian Heritage | 0 | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 46 | 48 | 50 | 144
  Multiple | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Determined by a Dermatologist to Have a Clinically Relevant Positive Outcome for Cutaneous Irritation After 21 Days of Product Use
Description: The clinically relevant positive outcome for cutaneous irritation was defined as the number of participants who experienced an increase in total cutaneous irritation score at Day 21 versus Baseline that was deemed clinically-relevant by the examiner. The dermatologist assessment of signs and symptoms of cutaneous irritation total score was calculated as the sum of the individual cutaneous response attributes (erythema, dryness, scaling, and edema). Each attribute was assessed on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Total possible score range was 0 to 12 where higher value indicated more cutaneous irritation.
Time Frame: Day 21
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 50 | 49 | 51
Participants | 1 | 0 | 0

2. Secondary Outcome: Number of Participants Determined by an Ophthalmologist to Have a Clinically Relevant Positive Outcome for Ocular Irritation After 21 Days of Product Use
Description: The clinically relevant positive outcome for ocular irritation was defined as the number of participants who experienced an increase in total ocular irritation score at Day 21 versus Baseline that was deemed clinically-relevant by the examiner. The ophthalmologist assessment of signs and symptoms of ocular irritation total score was calculated as the sum of the individual ocular response attributes (eczema of the eyelid, conjunctivitis, follicles, and chemosis conjunctivae). Each attribute was assessed on a scale with a score range of 0 to 3, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. Total possible score range was 0 to 12 where higher value indicated the most severe condition.
Time Frame: Day 21
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 50 | 49 | 51
Participants | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline (Prior to Any Product Application) in Participant Self-Assessment Scores of Signs and Symptoms of Cutaneous Irritation 1 to 2 Hours After First Product Application
Description: Participants were asked to self-assess any sensations of cutaneous discomfort for redness, dryness, stinging/burning, itching, and tightness each on separate 0-3 scale, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. These 5 separate assessments were summed to give an overall self-assessed total signs and symptoms of cutaneous irritation score ranging from 0-15. A high score indicates the most severe condition. Change from Baseline in total score at 1 to 2 hours = total cutaneous score at 1 to 2 hours minus total cutaneous score at Baseline. Negative values reflect improvement; a decrease in total score versus Baseline. This reflects a reduction in total signs and symptoms of cutaneous irritation versus Baseline. Positive values reflect worsening; an increase in total score versus Baseline. This reflects an increase in total signs and symptoms of cutaneous irritation versus Baseline. A zero change reflects no change in total score.
Time Frame: Baseline and 1 to 2 hours post first use
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 50 | 49 | 51
Participants
  Total score= -14 | 0 | 1 | 0
  Total score= -10 | 0 | 0 | 1
  Total score= -9 | 0 | 1 | 0
  Total score= -8.5 | 0 | 1 | 0
  Total score= -8 | 0 | 0 | 1
  Total score= -7.5 | 2 | 0 | 0
  Total score= -7 | 1 | 0 | 0
  Total score= -6 | 2 | 1 | 3
  Total score= -5.5 | 0 | 0 | 2
  Total score= -5 | 2 | 3 | 0
  Total score= -4.5 | 2 | 7 | 1
  Total score= -4 | 4 | 5 | 5
  Total score= -3.5 | 4 | 3 | 6
  Total score= -3 | 4 | 5 | 5
  Total score= -2.5 | 3 | 5 | 3
  Total score= -2 | 5 | 6 | 5
  Total score= -1.5 | 5 | 3 | 7
  Total score= -1 | 6 | 3 | 4
  Total score= -0.5 | 2 | 3 | 7
  Total score= 0 | 4 | 0 | 1
  Total score= 0.5 | 2 | 2 | 0
  Total score= 2 | 1 | 0 | 0
  Total score= 3 | 1 | 0 | 0

4. Secondary Outcome: Change From Baseline (Prior to Any Product Application) in Participant Self-Assessment Scores of Signs and Symptoms of Cutaneous Irritation After 21 Days of Product Use
Description: Participants were asked to self-assess any sensations of cutaneous discomfort for redness, dryness, stinging/burning, itching, and tightness each on separate 0-3 scale, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. These 5 separate assessments were summed to give an overall self-assessed total signs and symptoms of cutaneous irritation score ranging from 0-15. A high score indicates the most severe condition. Change from Baseline in total score at Day 21 = total cutaneous score at Day 21 minus total cutaneous score at Baseline. Negative values reflect improvement; a decrease in total score versus Baseline. This reflects a reduction in total signs and symptoms of cutaneous irritation versus Baseline. Positive values reflect worsening; an increase in total score versus Baseline. This reflects an increase in total signs and symptoms of cutaneous irritation versus Baseline. A zero change reflects no change in total score.
Time Frame: Baseline and Day 21
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 49 | 47 | 51
Participants
  Total score= -14 | 0 | 1 | 0
  Total score= -10.5 | 1 | 0 | 0
  Total score= -10 | 0 | 0 | 1
  Total score= -9 | 0 | 1 | 0
  Total score= -8.5 | 0 | 1 | 1
  Total score= -8 | 0 | 1 | 2
  Total score= -7.5 | 2 | 1 | 0
  Total score= -6.5 | 3 | 0 | 1
  Total score= -6 | 0 | 2 | 1
  Total score= -5.5 | 1 | 1 | 2
  Total score= -5 | 3 | 5 | 1
  Total score= -4.5 | 2 | 1 | 1
  Total score= -4 | 2 | 2 | 2
  Total score= -3.5 | 0 | 3 | 3
  Total score= -3 | 2 | 5 | 6
  Total score= -2.5 | 6 | 4 | 5
  Total score= -2 | 4 | 3 | 4
  Total score= -1.5 | 6 | 4 | 10
  Total score= -1 | 7 | 5 | 1
  Total score= -0.5 | 3 | 3 | 3
  Total score= 0 | 4 | 3 | 5
  Total score= 0.5 | 1 | 0 | 0
  Total score= 1 | 2 | 0 | 1
  Total score= 2 | 0 | 1 | 1

5. Secondary Outcome: Change From Baseline Prior to Any Product Application) in Participants Self-Assessment Scores of Signs and Symptoms of Ocular Irritation 1 to 2 Hours After First Product Application
Description: Participants were asked to self-assess any sensations of ocular discomfort for redness, dryness, stinging/burning, and itching each on separate 0-3 scale, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. These 5 separate assessments were summed to give an overall self-assessed total signs and symptoms of ocular discomfort score ranging from 0-12. A high score indicates the most severe condition. Change from Baseline in total score at 1 to 2 hours = total ocular score at 1 to 2 hours minus total ocular score at Baseline. Negative values reflect improvement; a decrease in total score versus Baseline. This reflects a reduction in total signs and symptoms of ocular irritation versus Baseline. Positive values reflect worsening; an increase in total score versus Baseline. This reflects an increase in total signs and symptoms of ocular irritation versus Baseline. A zero change reflects no change in total score.
Time Frame: Baseline and 1 to 2 hours post first use
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 50 | 49 | 51
Participants
  Total score= -3 | 2 | 1 | 0
  Total score= -2.5 | 0 | 2 | 1
  Total score= -2 | 1 | 2 | 0
  Total score= -1.5 | 1 | 1 | 2
  Total score= -1 | 2 | 4 | 6
  Total score= -0.5 | 7 | 7 | 4
  Total score= 0 | 37 | 32 | 35
  Total score= 0.5 | 0 | 0 | 2
  Total score= 1 | 0 | 0 | 1

6. Secondary Outcome: Change From Baseline (Prior to Any Product Application) in Participant Self-Assessment Scores of Signs and Symptoms of Ocular Irritation After 21 Days of Product Use
Description: Participants were asked to self-assess any sensations of ocular discomfort for redness, dryness, stinging/burning, and itching each on separate 0-3 scale, where 0=none, 0.5=very slight, 1=slight, 2=moderate, 3=severe. These 5 separate assessments were summed to give an overall self-assessed total signs and symptoms of ocular discomfort score ranging from 0-12. A high score indicates the most severe condition. Change from Baseline in total score at Day 21 = total ocular score at Day 21 minus total ocular score at Baseline. Negative values reflect improvement; a decrease in total score versus Baseline. This reflects a reduction in total signs and symptoms of ocular irritation versus Baseline. Positive values reflect worsening; an increase in total score versus Baseline. This reflects an increase in total signs and symptoms of ocular irritation versus Baseline. A zero change reflects no change in total score.
Time Frame: Baseline and Day 21
Population: Safety Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
Number analyzed (Participants) | 49 | 47 | 51
Participants
  Total score= -5 | 2 | 0 | 0
  Total score= -3 | 1 | 1 | 0
  Total score= -2.5 | 0 | 1 | 1
  Total score= -2 | 0 | 2 | 1
  Total score= -1.5 | 2 | 3 | 1
  Total score= -1 | 1 | 2 | 5
  Total score= -0.5 | 9 | 7 | 7
  Total score= 0 | 28 | 21 | 28
  Total score= 0.5 | 2 | 5 | 4
  Total score= 1 | 2 | 4 | 2
  Total score= 1.5 | 1 | 0 | 0
  Total score= 2.5 | 0 | 0 | 1
  Total score= 3 | 0 | 1 | 0
  Total score= 4.5 | 0 | 0 | 1
  Total score= 6 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening up to Final Visit (Day 21)
Description: Treatment-emergent Adverse Events (TEAEs) were defined as new Adverse Events (AEs) that occurred on or after the first study product application (if this date was missing, a suitable alternative was used). AEs with an onset date/time prior to the first study product application were considered as non-treatment emergent.
Arm/Group | Developmental Serum | Developmental Lotion | Developmental Cream
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49 | 0/51
Other Adverse Events (participants affected / at risk) | 5/50 | 6/49 | 4/51
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Developmental Serum (N=50) | Developmental Lotion (N=49) | Developmental Cream (N=51)
Headache (Nervous system disorders) | 2 | 3 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
NASAL MUCOSAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
EYE IRRITATION (Eye disorders) | 1 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04557371/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT04557371/SAP_001.pdf